CLINICAL TRIAL: NCT07241884
Title: SakuraBead Used as Resorbable Embolic for Plantar Fascia Embolization
Acronym: SURE-PF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CrannMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI580
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Plantar Fascitis; Heel Pain; Musculoskeletal Diseases
Keywords: Fasciitis; Musculoskeletal disease; Foot disease; Heel Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Fasciitis; Foot Diseases | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arterial Embolisation (Experimental): Temporary embolization using resorbable microspheres
  Interventions: Device: Arterial Embolization
- Shockwave (Active Comparator): Extracorporeal Shockwave Therapy (ESWT); a non-invasive therapeutic approach used to treat a variety of musculoskeletal conditions, including plantar fasciitis.
  Interventions: Device: Extracorporeal shockwave therapy

INTERVENTIONS:
Device: Arterial Embolization — Resorbable microspheres are delivered trans-arterially using a microcatheter or introducer sheath to the site of embolization where they will temporarily embolize the hypervascularity in the targeted region with preservation of normal arterial flow.
  Arms: Arterial Embolisation
Device: Extracorporeal shockwave therapy — Extracorporeal shockwave therapy (ESWT) is a treatment using acoustic pulses to treat plantar fasciitis.
  Arms: Shockwave

SUMMARY:
This is a prospective, single center, double arm, randomized, unmasked, First in Human study that aims to evaluate the safety and effectiveness of SakuraBead™ resorbable embolization microspheres in adult patients suffering from pain secondary to plantar fasciitis.

DETAILED DESCRIPTION:
To compare safety and efficacy of SakuraBead with shockwave therapy for the treatment of pain secondary to plantar fasciitis. Treatment will be performed on a total of approximately 45 patients who will be followed up for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able and willing to provide written informed consent, and
2. Age 18 to 75 years (inclusive), and
3. Clinical diagnosis of PF with proximal plantar fascia thickness greater than 4mm and areas of hypoechogenicity.

Exclusion Criteria:

1. Acute internal derangement of the foot including acute meniscal, ligament or bone injury, or
2. Sensory or motor neuropathy of the feet, or
3. Heel pain caused by stress fractures, nerve entrapment, or inflammatory conditions such as arthritis, gout, or bursitis, or
4. Prior surgical repair or plantar fascia rupture in the involved foot, or
5. Local infection in either foot, or
6. Contraindication to MRI, or
7. Active pregnancy as demonstrated by urine or serum β-hCG or lactating female
8. Unable to provide informed consent or comply with the conditions of the study, or
9. At the discretion of the Principal Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 3 Months
  Compare the proportion of responders between the Investigational procedure and Control.
Primary Safety Endpoint | 3 months
  Freedom from device or procedure-related serious adverse events (SAE) following the index procedure (proportions will be compared between Investigational procedure and Control).

CONTACTS AND LOCATIONS:
Locations (1):
- Nano Medical Clinic, Tashkent, Uzbekistan, Uzbekistan

IPD SHARING:
Plan to Share IPD: No